CLINICAL TRIAL: NCT03496259
Title: On-Q Pump vs Epidural for Postoperative Pain Control in Children Undergoing Oncologic Surgery
Brief Title: On-Q Pump vs Epidural for Postoperative Pain Control in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment, one of investigators left institution.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Bindi Naik-Mathuria, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-42606
Record Dates: First submitted 2018-03-30; First posted 2018-04-12 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain, on-Q pump, epidural, children
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, family and clinical care team (nurses, residents, physician assistants) will be blinded, as well as the research team collecting outcomes. The surgeons (including primary investigator) will not be blinded as will be placing the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-Q Group (Experimental): Patients in this group will have an On-Q pump placed at the end of the operation
  Interventions: Device: On-Q pump
- Epidural Group (Active Comparator): Patients in this group will have an epidural catheter placed at the end of the operation
  Interventions: Device: Epidural catheter

INTERVENTIONS:
Device: On-Q pump — Type of pain control device used
  Arms: On-Q Group
Device: Epidural catheter — Type of pain control device used
  Arms: Epidural Group

SUMMARY:
Open abdominal and pelvic surgery or thoracotomy (open chest surgery) is frequently performed for tumor excision in children. Post-operative pain management regimens are often at the discretions of the attending surgeon and may include opiods, patient administered analgesia (PCA), epidural catheters, subcutaneous analgesia catheters or NSAIDS to control incisional pain. Currently, both epidural or subcutaneous analgesia catheters (On-Q pumps) are commonly used for children undergoing these operations, at the discretion of the surgeon. There are no studies comparing these regimens in children. The purpose of this study is to compare postoperative pain control of the two strategies.

DETAILED DESCRIPTION:
The study design is a randomized, controlled trial to compare the effectiveness of on-q pump subcutaneous incisional analgesia to epidural analgesia for postoperative pain relief in children undergoing open abdominal, thoracic, or pelvic operations for oncologic purposes. The patient and treating team will be blinded to the pain control device. The primary outcome is additional narcotic usage for 3 post-operative days, and secondary outcomes are pain scores for 3 post-operative days, post-surgical day of ambulation, time to regular diet, infectious complications (UTI, wound infection or pneumonia), and hospital length of stay. Outcomes from both groups will be directly compared in order to determine whether one strategy provides more effective pain control with less complications than the other, or whether they are equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 5kg
* Age younger than 19 years of age
* Planned abdominal, pelvic or thoracic operation for an oncologic indication

Exclusion Criteria:

* Patients deemed inappropriate for placement of epidural by anesthesiologist
* Minimally invasive operation
* Biopsy through limited incision
* History of chronic narcotic or opioid use
* History of drug abuse

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Additional narcotic use | 3 days
  Mg of additional narcotics used for 3 post-operative days

SECONDARY OUTCOMES:
Pain scores | 3 days
  Visual analog scores provided by patients every 4 hours will be collected for 3 post-operative days
Days to ambulation | 0-5 days
  The first post-operative day that patients are ambulating outside the room will be noted
Days to initiation of regular diet | 0-5 days
  The first post-operative day of initiation of a regular diet will be noted
Development of postoperative infection | 0-5 days
  Infections (such as urinary tract infection, wound infection, or epidural site infection) will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Bindi Naik-Mathuria, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No